CLINICAL TRIAL: NCT04829604
Title: A Global, Phase 2 Study of ARX788 in HER2-positive Metastatic Breast Cancer Patients Who Were Previously Treated With T-DXd
Brief Title: ARX788 in HER2-positive, Metastatic Breast Cancer Subjects (ACE-Breast-03)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ambrx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Breast-03
Record Dates: First submitted 2021-03-18; First posted 2021-04-02 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: HER2 Positive Metastatic Breast Cancer
Keywords: HER2-postive; Breast cancer; Antibody drug; Metastatic; ARX788; HER2
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — ARX788; Immunoconjugates

STUDY DESIGN:
Intervention Model Description: One single arm, open label with intravenous infusion of ARX788 to assess the anticancer activity and safety of ARX788 in subjects with unresectable or metastatic human epidermal growth factor receptor 2 (HER2)-positive (HER2+) breast cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARX788 (Experimental): The investigational medicinal product (IMP), ARX788, will be administered every 3 weeks (Q3W) by intravenous (IV) infusion.
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — The active pharmaceutical ingredient in ARX788 is an antibody drug conjugate (ADC) consisting of a humanized anti-HER2 monoclonal antibody (mAb) (IgG1κ) covalently conjugated to two microtubule-disrupting payloads AS269
  Other Names: antibody drug conjugate (ADC)

SUMMARY:
A Global, Phase 2 Study of ARX788 in HER2-positive Metastatic Breast Cancer Patients who were previously treated with T-DXd

DETAILED DESCRIPTION:
A Global, Single Arm, Phase 2 Study of ARX788 in HER2-positive Metastatic Breast Cancer Patients who were previously treated with T-DXd. The ARX788 will be administered every 3 weeks (Q3W) intravenous (IV) infusion.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years and older
* Life expectancy ≥ 6 months
* Unresectable or metastatic breast cancer subjects
* Presence of at least one measurable lesion per RECIST v 1.1
* Subjects must have HER2 positive breast cancer per ASCO-CAP guidelines, documented in a CLIA lab pathology report
* Subjects must have had prior treatment with no more than 5 prior regimens of systemic treatment HER-2 targeting therapy or chemotherapy in the metastatic setting. One of these prior treatments must have been treatment with T-DXd.
* Subjects with stable brain metastases
* Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade ≤1 as per the NCI-CTCAE v 5.0, except alopecia, vitiligo, Grade 2 peripheral neuropathy, or endocrine toxicities that are stable on hormone replacement.
* Adequate organ functions
* Willing and able to understand and sign an informed consent inform and to comply with all aspects of the protocol

Key Exclusion Criteria:

Any subject who meets any of the following criteria is excluded from the study:

* History of allergic reactions to any component of ARX788.
* Prior history of interstitial lung disease, pneumonitis, or other clinically significant lung disease. Any requirement for supplemental oxygen.
* Any active ocular infections or chronic corneal disorders
* History of congestive heart failure, unstable angina pectoris, unstable atrial fibrillation, cardiac arrhythmia, or myocardial infarction within 6 months prior to enrollment
* Grade 3 to 4 peripheral neuropathy (NCI CTCAE v 5.0).
* History of unstable central nervous system (CNS) metastases
* Radiotherapy outside of the brain administered < 7 days prior to first dose of ARX788
* Current severe, uncontrolled systemic disease (eg, clinically significant cardiovascular, pulmonary, or metabolic diseases)
* Any uncontrollable intercurrent illness, infection (including subjects with active, symptomatic Covid-19 infections), or other conditions that could limit study compliance or interfere with assessments
* Exposure to any other investigational or commercial anticancer agents or therapies administered with the intention to treat malignancy within 14 days before the first dose of ARX788

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2021-10-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 2 years
  To evaluate the confirmed objective response rate (ORR) as determined by Investigator assessment based on Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) following treatment with ARX788.
  The ORR is defined as the number of subjects with a BOR of CR or PR divided by the number of response evaluable subjects.

SECONDARY OUTCOMES:
Duration of response (DOR) | 2 years
  DOR is defined as the time between the date of first response and the date of disease progression or death, whichever occurs first, will be computed for subjects with a BOR of CR or PR.
Best overall response (BOR) | 2 years
  BOR is defined as the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started)
Disease control rate (DCR) | 2 years
  DCR is defined as the proportion of complete response (CR), partial response (PR), and stable disease (SD) rates.
Overall survival (OS) | 2.5 years
  Overall survival (OS) is defined as the time from first dose of study therapy to the date of death (any cause). Subjects who are alive will be censored at the last known time that the subject was alive.
Progression-free survival (PFS) | 2 years
  PFS is defined as the time between date of first dose of study therapy and date of progression or death, whichever occurs first, will be computed for response evaluable subjects. Subjects will be censored at time of subsequent therapy
The number of subjects experiencing adverse event TEAEs | 2 years
  Patient safety and adverse events (AEs) will be evaluated using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.5.0. All AEs and serious adverse events (SAEs) will be assessed to determine the safety and tolerability of the treatment.
Maximum serum concentration (Cmax) for ARX788 | Cycle 1 and cycle 3
  Pharmacokinetic parameter maximum serum concentration (Cmax) for ARX788, ADC, ADA, total antibody, and pAF-AS269
Trough concentration (Ctrough) for ARX788 | Cycle 1 and cycle 3
  Pharmacokinetic parameter trough concentration (Ctrough) for ARX788, ADC, total antibody, and pAF-AS269
Area under the serum concentration-time curve (AUC) for ARX788 | Cycle 1 and cycle 3
  Pharmacokinetic parameter area under the serum concentration-time curve (AUC) for ARX788, ADC, total antibody, and pAF-AS269
Time to response (TTR) | Start of treatment to first objective confirmed BOR of CR or PR, assessed for approximately 2 years
  Time it takes for patient to respond to study treatment

OTHER OUTCOMES:
Evaluate Biomarker | 2 years
  To evaluate exploratory blood- and tissue-based biomarkers related to study drug response

CONTACTS AND LOCATIONS:
Overall Officials: Ambrx, Study Director — Ambrx, Inc.
Locations (31):
- United States (25):
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, San Francisco, California
  - Research Site, Whittier, California
  - Research Site, Athens, Georgia
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Louisville, Kentucky
  - Research Site, Silver Spring, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Camden, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Shirley, New York
  - Research Site, The Bronx, New York
  - Research Site, Portland, Oregon
  - Research Site, Tigard, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
- Australia (3):
  - Research Site, Frankston, Victoria
  - Research Site, Geelong, Victoria
  - Research Site, Nedlands, Western Australia
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Seongnam-si
  - Research Site, Seoul